CLINICAL TRIAL: NCT03068884
Title: Dopaminergic Contribution to Behavioural Flexibility as Modulated by Transcranial Direct-current Stimulation of the Dorsolateral Prefrontal Cortex
Brief Title: Dopamine Dorsolateral Prefrontal Cortex Behavioural Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SheffieldHallamAquili2017
Record Dates: First submitted 2017-02-21; First posted 2017-03-03 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Cognitive Change
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Tyrosine; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tdcs sham (Sham Comparator)
  Interventions: Dietary Supplement: L-Tyrosine; Dietary Supplement: Cellulose (placebo)
- Placebo (Placebo Comparator)
  Interventions: Device: Cathodal Transcranial direct current stimulation; Device: Transcranial direct current stimulation (sham)
- Tdcs cathodal (Experimental)
  Interventions: Dietary Supplement: L-Tyrosine; Dietary Supplement: Cellulose (placebo)
- Tyrosine (Experimental)
  Interventions: Device: Cathodal Transcranial direct current stimulation; Device: Transcranial direct current stimulation (sham)

INTERVENTIONS:
Device: Cathodal Transcranial direct current stimulation — Cathodal transcranial direct current stimulation over the dorsolateral prefrontal cortex
  Arms: Placebo; Tyrosine
Dietary Supplement: L-Tyrosine — Administration of 2 grams tyrosine
  Arms: Tdcs cathodal; Tdcs sham
Device: Transcranial direct current stimulation (sham) — Sham tDCS
  Arms: Placebo; Tyrosine
Dietary Supplement: Cellulose (placebo) — Administration of 2 grams cellulose
  Arms: Tdcs cathodal; Tdcs sham

SUMMARY:
Behavioural or cognitive flexibility (BF) is an essential ability which allows an organism to adaptively change responses in accordance with feedback of results. In humans, this ability is disrupted among those who suffer a variety of neurological and psychiatric conditions including Parkinson's disease, schizophrenia, addiction, obsessive compulsive disorder and autism. Additionally, there is evidence of substantial individual differences in BF within the healthy population.

Two known neurobiological mechanisms which relate to BF performance are variation in dopamine (DA) and serotonin (SE) function. One particular brain regions which has been heavily implicated in BF is the prefrontal cortex (PFC), with the dorsolateral PFC receiving a largely DA innervation and the dorsomedial PFC a SE input. Studies have demonstrated that damage to parts of PFC including the orbitofrontal cortex (OFC), for example, impairs reversal learning (a form of BF) whereas lesions of the dorsolateral PFC affect attentional set-shifting (another measure of BF).

In humans, putative augmentation of DA efflux via administration of the DA and norepinephrine precursor tyrosine has been shown to improve task-switching performance, and inhibitory control suggesting a causal role of DA in regulating BF. Similarly, putative depletion of serotonin neurotransmission via tryptophan depletion procedures has been shown to reduce the BOLD response during performance monitoring and increase perseverative behaviour.

One important strategy (in humans) to observe whether the PFC is causally involved in BF performance, is by reversible electrical stimulation of the PFC, so that PFC cells could be inhibited or excited while a participant is performing a BF task. In recent years, several laboratories have taken advantage of a relatively new technology known as transcranial direct current stimulation (tDCS) to study the relationship between brain function and behaviour. Using this technique, increases or decreases in cortical excitability are partly determined by the polarity of the stimulation; increases occur under the anode electrode whereas decreases occur under the negatively charged cathode.

Using this approach, several studies have shown that anodal and cathodal stimulation over the PFC can have a number of effects on BF performance, with general improvements during anodal stimulation and impairments during cathodal. If this is the case, one important step that remains to be understood is whether dopamine and serotonin are causally related to these outcomes when neurons of the dLPFC/dMPFC are either excited or inhibited via tDCS.

Thus, the specific novelty of this study rests in combining a psychopharmacological approach (i.e. tyrosine/tryptophan loading) with selective neuroanatomical (i.e. dorsolateral/dorsomedial prefrontal cortex) inhibition of cells via tDCS while participants are performing BF tasks. By doing so, we will be able to establish whether increased dopaminergic/serotonergic output to the PFC is a necessary requirement for BF performance.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years
* In good health
* Agrees to fast overnight prior to testing

Exclusion Criteria:

* Presence of cardiac, hepatic, renal, or neurological disorders
* Presence of damaged or diseased skin on your face and scalp, or a sensitive scalp
* A history of alcohol or drug addiction, or severe psychiatric illness
* Taking drugs which may lower seizure threshold (i.e. epilepsy)
* In a state of pregnancy
* Having slept less than 6 hours the night before testing
* A history of migraine or headaches
* A history of taking antidepressants
* A history of taking tyrosine supplements

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Wisconsin Card Sorting task | 2 hours for each of the four conditions
  Total Number of errors (e.g. 1-200)
Probabilistic reversal learning task | 2 hours for each of the four conditions
  Mean Errors per reversal (e.g. 1-20)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Aquili, Ph.D., Principal Investigator — Sheffield Hallam University
Locations (1):
- Psychology laboratories, Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No